CLINICAL TRIAL: NCT06318429
Title: Evaluation of the Effect of Stretching Exercises Applied to Diabetes Patients on Physiological Parameters and Compliance to Treatment: A Randomized Controlled Study
Brief Title: Effect of Stretching Exercises Applied to Diabetes Patients Physiological Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Gürcan Solmaz, Assistant Professor, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: diabet
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
Keywords: diabetes; exercise; blood sugar
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stretching exercise group (Experimental): stretching exercise group
  Interventions: Behavioral: stretching exercise group
- control group (No Intervention): control group

INTERVENTIONS:
Behavioral: stretching exercise group — stretching exercise group
  Arms: stretching exercise group

SUMMARY:
This research will be carried out as a pretest-posttest randomized controlled study to determine the effect of stretching exercises performed 2 days a week for 12 weeks for one hour each session on physiological parameters and treatment compliance in individuals with diabetes.

DETAILED DESCRIPTION:
This research will be carried out as a pretest-posttest randomized controlled study to determine the effect of stretching exercises performed 2 days a week for 12 weeks for one hour each session on physiological parameters and treatment compliance in individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Those who have been diagnosed with diabetes and have been on the same diabetes treatment for at least three months
3. Non-pregnant
4. Those who agreed to participate in the research
5. Those without any physical exercise disability

Exclusion Criteria:

1. Illiterate
2. Persons with severe mental disorders
3. Those who do not wish to answer the survey questions
4. Those who do not agree to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
blood sugar | 12 weeks
  fasting blood glucose measurement

CONTACTS AND LOCATIONS:
Locations (1):
- University of İstanbul-cerrahpaşa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solmaz G. The Effects of Yoga Practice on Glycemic Control and Self-Care Among Low Socioeconomic Status Women with Type 2 Diabetes: A Randomized Controlled Trial. Niger J Clin Pract. 2025 Oct 1;28(10):1121-1129. doi: 10.4103/njcp.njcp_491_25. Epub 2025 Oct 31. PMID 41307367